CLINICAL TRIAL: NCT00296517
Title: Clinical Evaluation of 323U66 SR in Patients With Depression - Placebo-controlled, Double-blind, Comparative Study in Patients With Depression Who Did Not Respond Sufficiently to Selective Serotonin Re-uptake Inhibitors
Brief Title: Study In Patients With Depression Not Responding to Selective Serotonin Re-uptake Inhibitors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK1102365
Record Dates: First submitted 2006-02-23; First posted 2006-02-27 (Estimated); Results first posted 2009-07-16 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2019-11

CONDITIONS: Depressive Disorder
Keywords: depression; double-blind; placebo-controlled; bupropion hydrochloride; SSRI; comparative study; non-responder
MeSH Terms: conditions — Depressive Disorder; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator): Subjects with Major Depressive Disorder who were randomised to placebo to match Bupropion SR during the treatment period.
  Interventions: Drug: Placebo
- Bupropion SR (Experimental): Subjects with Major Depressive Disorder who were randomized to take 100mg of Bupropion SR in the morning and placebo in the evening for one week. Week 2 subjects were given 100mg dose of Bupropion morning and evening. Weeks 3 thru 12 received 150mg dose morning and evening. Week 1=dose level 1, 100 mg. Week 2=dose level 2, 200 mg. Weeks 3 - 12=dose level 3, 300 mg.
  Interventions: Drug: 323U66 (Bupropion Hydrochloride Sustained Release)

INTERVENTIONS:
Drug: 323U66 (Bupropion Hydrochloride Sustained Release) — Subjects with Major Depressive Disorder who were randomized to take 100mg of Bupropion SR in the morning and placebo in the evening for one week. Week 2 subjects were given 100mg dose of Bupropion morning and evening. Weeks 3 thru 12 received 150mg dose morning and evening. Week 1=dose level 1, 100 mg. Week 2=dose level 2, 200 mg. Weeks 3 - 12=dose level 3, 300 mg.
  Arms: Bupropion SR
Drug: Placebo — Subjects with Major Depressive Disorder who were randomised to placebo to match Bupropion SR during the treatment period.
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the efficacy and safety in depressive patients who did not respond sufficiently to selective serotonin re-uptake inhibitors (SSRI).

ELIGIBILITY:
Inclusion criteria:

* [At the start of the pretreatment phase]
* Target disease: Patients diagnosed as having the following primary disease on the basis of DSM-IV-TR criteria.
* Major Depressive Disorder, Single Episode (296.2x) (excluding with psychotic features)
* Major Depressive Disorder, Recurrent (296.3x) (excluding with psychotic features)
* HAM-D (17 items) total score is >=16.
* Patients who have been treated with marketed paroxetine (Paxil®) at 20mg/day to 40mg/day for 4 weeks and more at the start of the pretreatment phase.
* Age: >=18 years old (at the time of informed consent) , <65 years old (at the start of treatment phase )
* Gender: Male or female.
* Inpatients or outpatients: Either
* Informed consent: The subject himself/herself must give written informed consent. However, if the subject is under 20 at the time of giving consent, both the subject himself/herself and his/her legally acceptable representative must give written informed consent.

[At the end of the pretreatment phase]

1. HAM-D (17 items) total score is ≥14.
2. Percentage of change from the start of the pretreatment phase in the HAM-D (17 items) total score is <50%

[At the start of the treatment phase]

1. HAM-D (17 items) total score is ≥14.
2. Percentage of change from the start of the pretreatment phase in the HAM-D (17 items) total score is <50%

Exclusion Criteria:

[At the start of the pre-treatment phase]

* Patients with a complication of glaucoma
* Patients concomitantly using a drug increasing the risk of bleeding and patients with bleeding tendency or predisposition to bleeding
* Patients with predisposition to seizure (who currently have or have a past history of seizure, febrile convulsive seizure in infancy, cerebral tumour, cerebrovascular disorder or head injury, who have a family history of idiopathic seizure, patients with diabetes who have been treated with oral hypoglycaemics or insulin, or who use drugs lowering the threshold of seizure).
* Patients who currently have or have a past history of the following disorders:
* Anorexia nervosa (DSM-IV-TR 307.1)
* Bulimia nervosa (DSM-IV-TR 307.51)
* Patients with a history of manic episode
* Patients with a past or current DSM- IV-TR diagnosis of schizophrenia or other psychotic disorder
* Patients with a current DSM-IV-TR Axis II diagnosis (e.g., antisocial or borderline personality disorder)
* Patients starting psychotherapy (except for supportive psychotherapy not aimed at therapeutic efficacy and unlikely to affect efficacy evaluation) and formal cognitive behaviour therapy within 5 weeks prior to the start of the pre-treatment phase
* Patients with a diagnosis of substance abuse (alcohol or drug) by the DSM-IV-TR criteria or with a diagnosis of substance dependence within 1 year prior to the start of the pre-treatment phase
* Patients who have received electroconvulsive therapy within 17 weeks prior to the start of the pre-treatment phase
* Patients who have taken MAO inhibitors (selegiline hydrochloride) within 2 weeks prior to the start of the pre-treatment phase
* Patients who have taken another investigational drug within 12 weeks prior to the start of the pre-treatment phase
* Female patients who are pregnant, possibly pregnant or are nursing, and those who want to become pregnant before 30 days after the last dose of the investigational product
* Patients who have attempted suicide within 17 weeks prior to the start of the pre-treatment phase, or patients for whom the score of suicide-related item No. 3 of HAM-D is >=3, or patients in whom the risk of suicide is judged to be high by the investigator (sub-investigator)
* Patients in whom the risk of homicide is judged to be high by the investigator (sub-investigator)
* Patients with a history of hypersensitivity to 323U66 and/or paroxetine
* Patients with serious cerebral disease
* Patients who have ECG or clinical evidence of any cardiac condition that the investigator (sub-investigator) feels may predispose the subject to ischemia or arrhythmia
* Patients with serious physical symptoms (i.e. cardiac/hepatic/renal disorder, hematopoietic disorder) The index of seriousness is Grade 3 of "Criteria for classification of seriousness of adverse drug reactions to pharmaceutical products, etc." (PAB/PSD No.80 in 1992).
* Patients with a history or complication of cancer or malignant tumour.
* Patients whose major depressive disorder is due to direct physiological effects of a general medical condition (for example, hypothyroidism, Parkinson's disease, chronic pain)
* Patients with systolic blood pressure of >=160 mmHg or diastolic blood pressure of >=100 mmHg
* Patients who are inappropriate for participating in the study in the judgement of the investigator (sub-investigator)

[At the start of the treatment phase]

1. Patients whose compliance of paroxetine during the pretreatment phase is less than 70%.
2. Patients who have ECG or clinical evidence of any cardiac condition that the investigator (sub-investigator) feels may predispose the subject to ischemia or arrhythmia
3. Patients with systolic blood pressure of >=160 mmHg or diastolic blood pressure of >=100 mmHg

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2006-01-19 (Actual); Primary Completion 2008-03-28 (Actual); Study Completion 2008-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (17):
- Japan (17):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Fukushima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Ishikawa
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Nara
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Tottori

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20096

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Pre-treatment period: Paroxetine 40 mg/day was administered for four weeks in subjects treated with marketed paroxetine between doses of 20 and 40 mg/day for four weeks or more prior to tapering pretreatment period.
  Tapering pretreatment period: Paroxetine was tapered down weekly by 10 mg/day in subjects who were progressed to treatment period.
Groups:
- Placebo: Subjects with Major Depressive Disorder who were randomized to placebo to match Bupropion SR during the treatment period.
- Bupropion SR: Subjects with Major Depressive Disorder who were randomized to take 100 mg of Bupropion SR in the morning and placebo in the evening for one week. Week 2 subjects were given 100 mg dose of Bupropion morning and evening. Weeks 3 through 12 received 150 mg dose morning and evening. Week 1 = dose level 1, 100 mg. Week 2 = dose level 2, 200 mg. Weeks 3 - 12 = dose level 3, 300 mg.
Period: Dose Level 1 - Week 1
Arm/Group | Placebo | Bupropion SR
Started | 159 | 166
Completed | 159 | 166
Not Completed | 0 | 0
Period: Dose Level 2 - Week 2
Arm/Group | Placebo | Bupropion SR
Started | 159 | 166
Completed | 157 | 161
Not Completed | 2 | 5
Not completed — Adverse Event | 1 | 5
Not completed — Withdrawal by Subject | 1 | 0
Period: Dose Level 3 - Weeks 3-12
Arm/Group | Placebo | Bupropion SR
Started | 157 | 161
Completed | 112 | 99
Not Completed | 45 | 62
Not completed — Adverse Event | 30 | 34
Not completed — Lack of Efficacy | 3 | 6
Not completed — Lost to Follow-up | 3 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 7 | 18
Not completed — Non - Compliance | 1 | 0
Not completed — Other | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Bupropion SR | Total
Number analyzed (Participants) | 157 | 165 | 322
Age, Continuous [Mean (Standard Deviation); unit: Years] — The Full Analysis Set (all subjects who entered the treatment phase, with the exception of those who did not take any investigational products during the treatment phase and those who did not meet the major eligibility criteria of Major Depressive Disorder or those with no valid post baseline assessment) for Baseline Characteristic measures.
  Years | 36.0 (8.91) | 36.8 (9.28) | 36.4 (9.10)
Sex: Female, Male [Count of Participants; unit: Participants] — The Full Analysis Set (all subjects who entered the treatment phase, with the exception of those who did not take any investigational products during the treatment phase and those who did not meet the major eligibility criteria of Major Depressive Disorder or those with no valid post baseline assessment) for Baseline Characteristic measures.
  Participants
    Female | 69 | 77 | 146
    Male | 88 | 88 | 176
Region of Enrollment [Number; unit: participants] — The Full Analysis Set (all subjects who entered the treatment phase, with the exception of those who did not take any investigational products during the treatment phase and those who did not meet the major eligibility criteria of Major Depressive Disorder or those with no valid post baseline assessment) for Baseline Characteristic measures.
  participants
    Japan | 157 | 165 | 322 (0) [0 to 0]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Hamilton Depression Scale (HAM-D 17 Items) Total Score
Description: The Hamilton Rating Scale for Depression contains 17 questions which detect change and measure illness severity. Individual items are rated on a scale of 0-4, 0-3, and 0-2 with total HAM-D score range from 0 (not ill) to 52 (severely ill).
Time Frame: Baseline and Week 12
Population: Full Analysis Set was all subjects who entered the treatment phase with the exception of those who did not take any investigational products during the treatment phase and those who did not meet the major eligibility criteria of Major Depressive Disorder or those with no valid post baseline assessment. Week 12/LOCF placebo = 155, Bupropion SR = 160
Measure: Mean (Standard Deviation); unit: Score in scale
Arm/Group | Placebo | Bupropion SR
Number analyzed (Participants) | 157 | 165
Score in scale
  Baseline | 19.8 (4.34) | 19.4 (4.39)
  Week 12 or Last Observation Carried Forward | 14.7 (8.89) | 14.6 (9.09)
  Change from Baseline | -5.1 (8.02) | -4.9 (8.34)
Statistical Analysis 1: Comparison: Placebo vs Bupropion SR; Null Hypothesis: The population mean change from baseline on HAM-D total score at Week 12 of the placebo group is equal to the population mean change from baseline on HAMD total score at Week 12 of the Bupropion hydrochloride sustained release group; Test type: Superiority or Other; p = 0.805, ANOVA; Mean Difference (Net) = 0.2, 95% CI [-1.6 to 2.0]

2. Secondary Outcome: Hamilton Depression Scale (HAM-D 17 Items) Total Score
Description: as for outcome 1
Time Frame: Week 8 and Week 12
Population: Full Analysis Set. Week 8 Last Observation Carried Forward: placebo = 152, Bupropion = 160, Week 8 Observed Cases: placebo = 113, Bupropion = 106, Week 12 Observed Cases: placebo = 111, Bupropion = 98
Measure: Mean (Standard Deviation); unit: Score in scale
Arm/Group | Placebo | Bupropion SR
Number analyzed (Participants) | 157 | 165
Score in scale
  Week 8 Mean - Last Observation Carried Forward | 15.8 (8.04) | 15.4 (8.32)
  Week 8 Mean - Observed Cases | 13.3 (6.74) | 12.1 (6.28)
  Week 12 Mean - Observed Cases | 11.3 (7.09) | 10.3 (6.83)

3. Secondary Outcome: Change From Baseline in the Hamilton Depression Scale (HAM-D 17 Items) Total Score at Week 8 and Total Score at Week 12
Description: as for outcome 1
Time Frame: Baseline to Week 8 and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score in a scale
Arm/Group | Placebo | Bupropion SR
Number analyzed (Participants) | 157 | 165
Score in a scale
  Week 8 Mean - Last Observation Carried Forward | -4.1 (7.07) | -4.0 (7.60)
  Week 8 Mean - Observed Cases | -6.4 (5.77) | -7.4 (5.75)
  Week 12 Mean - Observed Cases | -8.3 (6.38) | -9.2 (5.98)

4. Secondary Outcome: Percentage of Change From Baseline of the Hamilton Depression (HAM-D 17 Items) Total Score at Weeks 8 and 12.
Description: as for outcome 1
Time Frame: Baseline to Week 8 and Week 12
Population: Full Analysis Set. Week 8 Last Observation Carried Forward: placebo = 152, Bupropion = 160, Week 8 Observed Cases: placebo = 113, Bupropion = 106, Week 12 Last Observation Carried Forward: placebo = 155, Bupropion = 160 Week 12 Observed Cases: placebo = 111, Bupropion = 98
Measure: Mean (Standard Deviation); unit: Percent Change in score
Arm/Group | Placebo | Bupropion SR
Number analyzed (Participants) | 157 | 165
Percent Change in score
  Week 8 Mean - Last Observation Carried Forward | -21.0 (37.31) | -20.8 (38.87)
  Week 8 Mean - Observed Cases | -33.2 (30.51) | -38.2 (28.68)
  Week 12 Mean - Last Observation Carried Forward | -26.5 (41.65) | -25.5 (43.05)
  Week 12 Mean - Observed Cases | -43.0 (32.51) | -48.4 (29.96)

5. Secondary Outcome: Percentage of Responders Based on Hamilton Depression (HAM-D 17 Items) Scale Total Score at Weeks 8 and 12
Description: The Hamilton Rating Scale for Depression contains 17 questions which detect change and measure illness severity. Individual items are rated on a scale of 0-4, 0-3, and 0-2 with total HAM-D score range from 0 (not ill) to 52 (severely ill). Responders are defined as subjects with 50% or greater reduction from baseline in HAM-D total score.
Time Frame: Baseline to Week 8 and Week 12
Population: Full Analysis Set. Week 8 Last Observation Carried Forward: placebo = 152, Bupropion = 160, Week 8 Observed Cases: placebo = 113, Bupropion = 106, Week 12 Last Observation Carried Forward: placebo = 155, Bupropion = 160, Week 12 Observed Cases: placebo = 111, Bupropion = 98
Measure: Mean (95% Confidence Interval); unit: Percentage of Responders
Arm/Group | Placebo | Bupropion SR
Number analyzed (Participants) | 157 | 165
Percentage of Responders
  Week 8 Mean Last Observation Carried Forward | 24 [17.8 to 32.0] | 26 [19.1 to 33.1]
  Week 8 Mean Observed Cases | 31 [22.6 to 40.4] | 38 [28.5 to 47.7]
  Week 12 Mean Last Observation Carried Forward | 37 [29.8 to 45.5] | 38 [30.6 to 46.1]
  Week 12 Mean Observed Cases | 50 [40.8 to 60.1] | 59 [48.8 to 69.0]

6. Secondary Outcome: Percentage of Remitters Based on Hamilton Depression (HAM-D 17 Items) Scale Total Score at Weeks 8 and 12
Description: The Hamilton Rating Scale for Depression contains 17 questions which detect change and measure illness severity. Individual items are rated on a scale of 0-4, 0-3, and 0-2 with total HAM-D score range from 0 (not ill) to 52 (severely ill). Remitters are defined as subjects with HAM-D total score ≤ 7.
Time Frame: Baseline to Week 8 and Week 12
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: Percentage of Remitters
Arm/Group | Placebo | Bupropion SR
Number analyzed (Participants) | 157 | 165
Percentage of Remitters
  Week 8 Mean Last Observation Carried Forward | 18 [12.0 to 24.8] | 18 [12.5 to 25.0]
  Week 8 Mean Observed Cases | 22 [14.9 to 30.9] | 26 [18.3 to 35.9]
  Week 12 Mean Last Observation Carried Forward | 25 [18.5 to 32.8] | 24 [17.4 to 31.1]
  Week 12 Mean Observed Cases | 33 [24.7 to 42.9] | 38 [28.2 to 48.1]

7. Secondary Outcome: Change From Baseline in Each Item of the Hamilton Depression Scale (HAM-D 17 Items) Score at Weeks 8 and 12
Description: The Hamilton Rating Scale for Depression contains 17 questions which detect change and measure illness severity. Individual items are rated on a scale of 0-4, 0-3, and 0-2, with total HAM-D scores ranging from 0 (not ill) to 54 (severely ill).
Time Frame: Baseline to Week 8 and Week 12
Population: Full Analysis Set. Week 8 Last Observation Carried Forward (LOCF): placebo=152, Bupropion=160; Week 12 LOCF: placebo=155, Bupropion=160. Gastrointestinal, GI.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Bupropion SR
Number analyzed (Participants) | 157 | 165
points on a scale
  Depressed Mood, Week 8 Mean LOCF | -0.5 (1.07) | -0.5 (1.20)
  Depressed Mood, Week 12 Mean LOCF | -0.6 (1.17) | -0.6 (1.30)
  Feelings of Guilt, Week 8 Mean LOCF | -0.3 (0.91) | -0.3 (0.75)
  Feelings of Guilt, Week 12 Mean LOCF | -0.3 (0.90) | -0.4 (0.77)
  Suicide, Week 8 Mean LOCF | -0.1 (0.82) | -0.1 (0.73)
  Suicide, Week 12 Mean LOCF | -0.1 (0.82) | -0.1 (0.72)
  Insomnia Early, Week 8 Mean LOCF | -0.3 (0.83) | -0.3 (0.82)
  Insomnia Early, Week 12 Mean LOCF | -0.4 (0.85) | -0.3 (0.89)
  Insomnia Middle, Week 8 Mean LOCF | -0.4 (0.87) | -0.3 (0.73)
  Insomnia Middle, Week 12 Mean LOCF | -0.4 (0.91) | -0.3 (0.79)
  Insomnia Late, Week 8 Mean LOCF | -0.3 (0.87) | -0.3 (0.78)
  Insomnia Late, Week 12 Mean LOCF | -0.3 (0.91) | -0.4 (0.88)
  Work and Activities, Week 8 Mean LOCF | -0.4 (0.93) | -0.4 (1.18)
  Work and Activities, Week 12 Mean LOCF | -0.6 (1.13) | -0.5 (1.35)
  Retardation, Week 8 Mean LOCF | -0.2 (0.69) | -0.2 (0.68)
  Retardation, Week 12 Mean LOCF | -0.3 (0.78) | -0.3 (0.73)
  Agitation, Week 8 Mean LOCF | -0.2 (0.68) | -0.2 (0.77)
  Agitation, Week 12 Mean LOCF | -0.3 (0.77) | -0.2 (0.77)
  Anxiety Psychic, Week 8 Mean LOCF | -0.3 (1.16) | -0.4 (1.10)
  Anxiety Psychic, Week 12 Mean LOCF | -0.5 (1.26) | -0.5 (1.19)
  Anxiety Somatic, Week 8 Mean LOCF | -0.2 (0.88) | -0.3 (0.92)
  Anxiety Somatic, Week 12 Mean LOCF | -0.3 (0.89) | -0.4 (0.99)
  Somatic Symptoms GI, Week 8 Mean LOCF | -0.1 (0.61) | 0.0 (0.74)
  Somatic Symptoms GI, Week 12 Mean LOCF | -0.1 (0.64) | -0.0 (0.80)
  Somatic Symptoms General, Week 8 Mean LOCF | -0.2 (0.65) | -0.2 (0.69)
  Somatic Symptoms General, Week 12 Mean LOCF | -0.2 (0.71) | -0.3 (0.71)
  Genital Symptoms, Week 8 Mean LOCF | -0.2 (0.58) | -0.2 (0.62)
  Genital Symptoms, Week 12 Mean LOCF | -0.2 (0.66) | -0.3 (0.71)
  Hypochondriasis, Week 8 Mean LOCF | -0.2 (0.77) | -0.1 (0.84)
  Hypochondriasis, Week 12 Mean LOCF | -0.3 (0.78) | -0.2 (0.89)
  Loss of Weight by History, Week 8 Mean LOCF | -0.1 (0.60) | -0.0 (0.58)
  Loss of Weight by History, Week 12 Mean LOCF | -0.1 (0.63) | 0.0 (0.64)
  Insight, Week 8 Mean LOCF | -0.1 (0.34) | -0.1 (0.41)
  Insight, Week 12 Mean LOCF | -0.1 (0.38) | -0.1 (0.45)

8. Secondary Outcome: Percentage of Change From Baseline in Each Item of the Hamilton Depression Scale (HAM-D 17 Items) Score at Weeks 8 and 12
Description: as for outcome 7
Time Frame: Baseline to Week 8 and Week 12
Population: Full Analysis Set. Last Observation Carried Forward, LOCF; Gastrointestinal, GI; Somatic, Som.; General, Gen.; Week, W.
Measure: Mean (Standard Deviation); unit: percent change in score
Arm/Group | Placebo | Bupropion SR
Number analyzed (Participants) | 157 | 165
percent change in score
  Depressed Mood, Week 8 Mean LOCF, n=152, 158 | -17.7 (60.38) | -18.5 (62.38)
  Depressed Mood, Week 12 Mean LOCF, n=155, 158 | -25.9 (62.78) | -22.2 (68.41)
  Feelings of Guilt, Week 8 Mean LOCF, n=128, 131 | -24.9 (55.10) | -25.8 (52.83)
  Feelings of Guilt, Week 12 Mean LOCF, n=129, 131 | -30.7 (56.34) | -30.8 (53.61)
  Suicide, Week 8 Mean LOCF, n=79, 75 | -34.2 (60.20) | -26.7 (70.87)
  Suicide, Week 12 Mean LOCF, n=80, 75 | -37.5 (56.53) | -26.0 (74.14)
  Insomnia Early, Week 8 Mean LOCF, n=112, 119 | -34.8 (53.20) | -29.8 (54.59)
  Insomnia Early, Week 12 Mean LOCF, n=114, 119 | -42.5 (53.73) | -31.9 (58.49)
  Insomnia Middle, Week 8 Mean LOCF, n=119, 124 | -42.0 (53.28) | -32.3 (51.48)
  Insomnia Middle, Week 12 Mean LOCF, n=122, 124 | -48.4 (54.90) | -37.1 (54.43)
  Insomnia Late, Week 8 Mean LOCF, n=109, 117 | -39.9 (56.43) | -31.6 (54.38)
  Insomnia Late, Week 12 Mean LOCF, n=110, 117 | -43.2 (61.88) | -37.2 (62.34)
  Work and Activities, Week 8 Mean LOCF, n=151, 156 | -16.6 (43.93) | -15.3 (55.66)
  Work and Activities, Week 12 Mean LOCF, n=154, 156 | -23.3 (47.61) | -19.4 (62.51)
  Retardation, Week 8 Mean LOCF, n=114, 124 | -28.4 (58.70) | -31.0 (53.19)
  Retardation, Week 12 Mean LOCF, n=117, 124 | -32.5 (63.08) | -38.3 (56.71)
  Agitation, Week 8 Mean LOCF, n=87, 99 | -38.7 (61.87) | -44.9 (60.40)
  Agitation, Week 12 Mean LOCF, n=89, 99 | -51.1 (64.83) | -44.9 (63.28)
  Anxiety Psychic, Week 8 Mean LOCF, n=146, 151 | -14.0 (58.25) | -17.9 (55.14)
  Anxiety Psychic, Week 12 Mean LOCF, n=148, 151 | -19.1 (62.70) | -21.0 (66.45)
  Anxiety Somatic, Week 8 Mean LOCF, n=144, 155 | -9.5 (57.89) | -13.9 (60.12)
  Anxiety Somatic, Week 12 Mean LOCF, n=147, 155 | -13.7 (59.35) | -17.7 (63.07)
  Somatic Symptoms GI, Week 8 Mean LOCF, n=95, 93 | -30.5 (56.16) | -25.8 (63.68)
  Somatic Symptoms GI, Week 12 Mean LOCF, n=97, 93 | -23.7 (62.12) | -34.9 (65.02)
  Somatic Symptoms Gen., Week 8 Mean LOCF, n=146,152 | -13.4 (50.61) | -18.8 (48.08)
  Som. Symptoms Gen., Week 12 Mean LOCF, n=149, 152 | -15.8 (54.55) | -23.7 (51.13)
  Genital Symptoms, Week 8 Mean LOCF, n=115, 129 | -15.2 (45.97) | -21.7 (45.86)
  Genital Symptoms, Week 12 Mean LOCF, n=118, 129 | -16.5 (51.50) | -29.5 (50.24)
  Hypochondriasis, Week 8 Mean LOCF, n=93, 102 | -34.6 (55.78) | -28.3 (63.70)
  Hypochondriasis, Week 12 Mean LOCF, n=95, 102 | -38.6 (56.82) | -38.1 (66.27)
  Loss of Weight by Hist., W 8 Mean LOCF, n=32, 26 | -60.9 (45.32) | -51.9 (57.41)
  Loss of Weight by Hist., W 12 Mean LOCF, n=34, 26 | -58.8 (48.42) | -57.7 (57.78)
  Insight, Week 8 Mean LOCF, n=48, 51 | -27.1 (44.91) | -41.2 (49.71)
  Insight, Week 12 Mean LOCF, n=49, 51 | -36.7 (48.71) | -47.1 (50.41)

9. Secondary Outcome: Change From Baseline in Clinical Global Impressions - Severity of Illness (CGI-S) Scale at Weeks 1, 2, 3, 4, and 8 and 12
Description: The 7-point Clinical Global Impressions-Severity of Illness Scale (CGI-S) measures the severity of psychiatric symptoms. The following scores can be given: 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; 7 = among the most extremely ill patients.
Time Frame: Baseline to Weeks 1, 2, 3, 4, 8, and 12
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Points on scale
Arm/Group | Placebo | Bupropion SR
Number analyzed (Participants) | 157 | 165
Points on scale
  Week 1 Mean LOCF, n=157, 165 | -0.0 (0.45) | 0.0 (0.51)
  Week 1 Mean OC, n=139, 143 | -0.1 (0.40) | -0.0 (0.45)
  Week 2 Mean LOCF, n=157, 165 | -0.1 (0.63) | -0.1 (0.71)
  Week 2 Mean OC, n=134, 132 | -0.2 (0.59) | -0.3 (0.66)
  Week 3 Mean LOCF, n=157, 165 | -0.2 (0.71) | -0.2 (0.73)
  Week 3 Mean OC, n=130, 127 | -0.3 (0.61) | -0.4 (0.65)
  Week 4 Mean LOCF, n=157, 165 | -0.2 (0.76) | -0.2 (0.83)
  Week 4 Mean OC, n=127, 116 | -0.4 (0.65) | -0.4 (0.77)
  Week 8 Mean LOCF, n=157, 164 | -0.5 (1.02) | -0.5 (1.01)
  Week 8 Mean OC, n=113, 106 | -0.7 (0.87) | -0.9 (0.85)
  Week 12 Mean LOCF, n=157, 163 | -0.6 (1.12) | -0.6 (1.15)
  Week 12 Mean OC, n=111, 98 | -0.9 (0.90) | -1.1 (0.98)

10. Secondary Outcome: Percentage of Responders Based on the Clinical Global Impression - Global Improvement (CGI-I) Scale at Weeks 8 and 12
Description: The CGI-I assesses the investigator's impression of the patient's current illness. The time span is the week before the rating and the score ranges from 1 (very much improved) to 7 (very much worse). Responders are subjects that have a score of 1 (very much improved) or 2 (much improved) on the CGI-I.
Time Frame: Baseline to Week 8 and Week 12
Population: Full Analysis set. Week 8 Last Observation Carried Forward: placebo = 153, Bupropion = 159; Week 8 Observed Cases: placebo = 113, Bupropion = 106; Week 12 Last Observation Carried Forward: placebo = 156, Bupropion = 158; Week 12 Observed Cases: placebo = 111, Bupropion = 98
Measure: Mean (95% Confidence Interval); unit: Percentage of Responders
Arm/Group | Placebo | Bupropion SR
Number analyzed (Participants) | 157 | 165
Percentage of Responders
  Week 8 Mean Last Observation Carried Forward | 33 [25.9 to 41.4] | 38 [30.8 to 46.4]
  Week 8 Mean Observed Cases | 42 [32.4 to 51.2] | 57 [46.6 to 66.2]
  Week 12 Mean Last Observation Carried Forward | 44 [35.7 to 51.8] | 48 [40.1 to 56.2]
  Week 12 Mean Observed Cases | 57 [47.0 to 66.1] | 73 [63.6 to 81.9]

11. Secondary Outcome: Study Continuation Rate as Assessed by the Number of Participants at Risk at Week 12
Description: Kaplan-Meier estimates were calculated using event or censoring and time to event or censoring. Participants at risk refers to participants with either a censoring or event time beyond the time point of interest (Week 12).
Time Frame: Week 12
Population: Full analysis set. Participants at risk refers to participants with either a censoring or event time beyond the time point of interest (Week 12).
Measure: Number; unit: participants
Arm/Group | Placebo | Bupropion SR
Number analyzed (Participants) | 157 | 165
participants
  Participants at risk | 102 | 90
  Participants not at risk | 55 | 75
Statistical Analysis 1: Comparison: Placebo vs Bupropion SR; Test type: Superiority or Other; p = 0.036, Log Rank

12. Secondary Outcome: Safety: Adverse Events by Organ System Class, Intensity, and Frequency
Description: Assessment of intensity was based on investigators/subinvestigator's clinical judgement per protocol instructions: Mild event, easily tolerated, with minimal discomfort and not interfering with Activities of Daily Living (ADLs); moderate event, with discomfort that interferes with ADLs; severe event, prevents ADLs.
Time Frame: Baseline to Week 12
Population: Safety population: comprised of participants who took at least one dose of the treatment period investigational product. The number of participants analyzed for this outcome measure represents the total number of events at each intensity.
Measure: Number; unit: Number of events
Arm/Group | Placebo | Bupropion SR
Number analyzed (Participants) | 159 | 166
Number of events
  Nervous System Disorders (NSD) - Any Event, mild | 32 | 31
  NSD - Any Event, moderate | 8 | 16
  NSD - Any Event, severe | 1 | 3
  NSD - Dizziness, mild | 11 | 8
  NSD - Dizziness, moderate | 4 | 8
  NSD - Dizziness, severe | 1 | 0
  NSD - Headache, mild | 6 | 8
  NSD - Headache, moderate | 3 | 6
  NSD - Headache, severe | 0 | 1
  NSD - Somnolence, mild | 10 | 8
  NSD - Somnolence, moderate | 0 | 0
  NSD - Somnolence, severe | 0 | 0
  NSD - Hypoesthesia, mild | 5 | 1
  NSD - Hypoesthesia, moderate | 1 | 0
  NSD - Hypoesthesia, severe | 0 | 0
  NSD - Dysgeusia, mild | 0 | 4
  NSD - Dysgeusia, moderate | 0 | 1
  NSD - Dysgeusia, severe | 0 | 0
  NSD - Depressed Level of Consciousness, mild | 0 | 1
  NSD - Depressed Level of Consciousness, moderate | 0 | 2
  NSD - Depressed Level of Consciousness, severe | 0 | 1
  NSD - Tremor, mild | 0 | 4
  NSD - Tremor, moderate | 0 | 0
  NSD - Tremor, severe | 0 | 0
  NSD - Convulsion, mild | 0 | 0
  NSD - Convulsion, moderate | 0 | 1
  NSD - Convulsion, severe | 0 | 1
  NSD - Dizziness postural, mild | 0 | 1
  NSD - Dizziness postural, moderate | 1 | 0
  NSD - Dizziness postural, severe | 0 | 0
  NSD - Dysesthesia, mild | 0 | 0
  NSD - Dysesthesia, moderate | 1 | 1
  NSD - Dysesthesia, severe | 0 | 0
  NSD - Parosmia, mild | 2 | 0
  NSD - Parosmia, moderate | 0 | 0
  NSD - Parosmia, severe | 0 | 0
  NSD - Akathisia, mild | 0 | 0
  NSD - Akathisia, moderate | 1 | 0
  NSD - Akathisia, severe | 0 | 0
  NSD - Anterograde Amnesia, mild | 1 | 0
  NSD - Anterograde Amnesia, moderate | 0 | 0
  NSD - Anterograde Amnesia, severe | 0 | 0
  NSD - Dysarthria, mild | 1 | 0
  NSD - Dysarthria, moderate | 0 | 0
  NSD - Dysarthria, severe | 0 | 0
  NSD - Head discomfort, mild | 1 | 0
  NSD - Head discomfort, moderate | 0 | 0
  NSD - Head discomfort, severe | 0 | 0
  NSD - Hyperesthesia, mild | 0 | 1
  NSD - Hyperesthesia, moderate | 0 | 0
  NSD - Hyperesthesia, severe | 0 | 0
  NSD - Loss of consciousness, mild | 0 | 1
  NSD - Loss of consciousness, moderate | 0 | 0
  NSD - Loss of consciousness, severe | 0 | 0
  NSD - Paraesthesia, mild | 0 | 1
  NSD - Paraesthesia, moderate | 0 | 0
  NSD - Paraesthesia, severe | 0 | 0
  Gastrointestinal Disorders (GID)-Any Event, mild | 28 | 32
  GID - Any Event, moderate | 15 | 14
  GID - Any Event, severe | 1 | 0
  GID - Nausea, mild | 12 | 16
  GID - Nausea, moderate | 8 | 10
  GID - Nausea, severe | 1 | 0
  GID - Diarrhea, mild | 6 | 6
  GID - Diarrhea, moderate | 3 | 1
  GID - Diarrhea, severe | 0 | 0
  GID - Vomiting, mild | 4 | 5
  GID - Vomiting, moderate | 4 | 2
  GID - Vomiting, severe | 0 | 0
  GID - Abdominal Pain upper, mild | 0 | 3
  GID - Abdominal Pain upper, moderate | 1 | 2
  GID - Abdominal Pain upper, severe | 0 | 0
  GID - Stomach Discomfort, mild | 2 | 3
  GID - Stomach Discomfort, moderate | 1 | 0
  GID - Stomach Discomfort, severe | 0 | 0
  GID - Constipation, mild | 5 | 0
  GID - Constipation, moderate | 0 | 0
  GID - Constipation, severe | 0 | 0
  GID - Abdominal Pain, mild | 1 | 3
  GID - Abdominal Pain, moderate | 0 | 0
  GID - Abdominal Pain, severe | 0 | 0
  GID - Stomatitis, mild | 1 | 2
  GID - Stomatitis, moderate | 0 | 1
  GID - Stomatitis, severe | 0 | 0
  GID - Toothache, mild | 2 | 0
  GID - Toothache, moderate | 1 | 0
  GID - Toothache, severe | 0 | 0
  GID - Abdominal Distension, mild | 0 | 2
  GID - Abdominal Distension, moderate | 0 | 0
  GID - Abdominal Distension, severe | 0 | 0
  GID - Gastritis, mild | 1 | 1
  GID - Gastritis, moderate | 0 | 0
  GID - Gastritis, severe | 0 | 0
  GID - Hypoesthesia oral, mild | 1 | 1
  GID - Hypoesthesia oral, moderate | 0 | 0
  GID - Hypoesthesia oral, severe | 0 | 0
  GID - Melaena, mild | 1 | 1
  GID - Melaena, moderate | 0 | 0
  GID - Melaena, severe | 0 | 0
  GID - Abdominal Pain Lower, mild | 0 | 0
  GID - Abdominal Pain Lower, moderate | 0 | 1
  GID - Abdominal Pain Lower, severe | 0 | 0
  GID - Dyspepsia, mild | 0 | 0
  GID - Dyspepsia, moderate | 1 | 0
  GID - Dyspepsia, severe | 0 | 0
  GID - Gingival Swelling, mild | 1 | 0
  GID - Gingival Swelling, moderate | 0 | 0
  GID - Gingival Swelling, severe | 0 | 0
  Infections and Infestations (INF)-Any Event, mild | 38 | 30
  INF - Any Event, moderate | 3 | 4
  INF - Any Event, severe | 0 | 0
  INF - Nasopharyngitis, mild | 31 | 24
  INF - Nasopharyngitis, moderate | 0 | 4
  INF - Nasopharyngitis, severe | 0 | 0
  INF - Gastrointestinal infection, mild | 3 | 3
  INF - Gastrointestinal infection, moderate | 0 | 0
  INF - Gastrointestinal infection, severe | 0 | 0
  INF - Bronchitis acute, mild | 0 | 3
  INF - Bronchitis acute, moderate | 0 | 0
  INF - Bronchitis acute, severe | 0 | 0
  INF - Bronchitis, mild | 1 | 0
  INF - Bronchitis, moderate | 1 | 0
  INF - Bronchitis, severe | 0 | 0
  INF - Gastroenteritis, mild | 1 | 0
  INF - Gastroenteritis, moderate | 1 | 0
  INF - Gastroenteritis, severe | 0 | 0
  INF - Enteritis Infectious, mild | 1 | 0
  INF - Enteritis Infectious, moderate | 0 | 0
  INF - Enteritis Infectious, severe | 0 | 0
  INF - Gastroenteritis viral, mild | 0 | 0
  INF - Gastroenteritis viral, moderate | 1 | 0
  INF - Gastroenteritis viral, severe | 0 | 0
  INF - Otitis Externa, mild | 1 | 0
  INF - Otitis Externa, moderate | 0 | 0
  INF - Otitis Externa, severe | 0 | 0
  INF - Purulence, mild | 1 | 0
  INF - Purulence, moderate | 0 | 0
  INF - Purulence, severe | 0 | 0
  INF - Rhinitis, mild | 0 | 1
  INF - Rhinitis, moderate | 0 | 0
  INF - Rhinitis, severe | 0 | 0
  INF - Vaginal Candidiasis, mild | 1 | 0
  INF - Vaginal Candidiasis, moderate | 0 | 0
  INF - Vaginal Candidiasis, severe | 0 | 0
  Psychiatric Disorders (PsyDO) - Any Event, mild | 8 | 10
  PsyDO - Any Event, moderate | 13 | 14
  PsyDO - Any Event, severe | 7 | 5
  PsyDO - Depression, mild | 2 | 2
  PsyDO - Depression, moderate | 11 | 9
  PsyDO - Depression, severe | 7 | 3
  PsyDO - Insomnia, mild | 0 | 4
  PsyDO - Insomnia, moderate | 1 | 1
  PsyDO - Insomnia, severe | 0 | 0
  PsyDO - Mood altered, mild | 3 | 2
  PsyDO - Mood altered, moderate | 0 | 1
  PsyDO - Mood altered, severe | 0 | 0
  PsyDO - Mania, mild | 0 | 0
  PsyDO - Mania, moderate | 1 | 0
  PsyDO - Mania, severe | 0 | 1
  PsyDO - Anxiety, mild | 1 | 0
  PsyDO - Anxiety, moderate | 0 | 0
  PsyDO - Anxiety, severe | 0 | 0
  PsyDO - Bipolar Disorder, mild | 0 | 0
  PsyDO - Bipolar Disorder, moderate | 0 | 0
  PsyDO - Bipolar Disorder, severe | 0 | 1
  PsyDO - Bruxism, mild | 0 | 1
  PsyDO - Bruxism, moderate | 0 | 0
  PsyDO - Bruxism, severe | 0 | 0
  PsyDO - Delerium, mild | 0 | 1
  PsyDO - Delerium, moderate | 0 | 0
  PsyDO - Delerium, severe | 0 | 0
  PsyDO - Depression suicidal, mild | 0 | 0
  PsyDO - Depression suicidal, moderate | 0 | 1
  PsyDO - Depression suicidal, severe | 0 | 0
  PsyDO - Dysphoria, mild | 0 | 1
  PsyDO - Dysphoria, moderate | 0 | 0
  PsyDO - Dysphoria, severe | 0 | 0
  PsyDO - Early morning awakening, mild | 0 | 0
  PsyDO - Early morning awakening, moderate | 0 | 1
  PsyDO - Early morning awakening, severe | 0 | 0
  PsyDO - Hallucination, mild | 0 | 1
  PsyDO - Hallucination, moderate | 0 | 0
  PsyDO - Hallucination, severe | 0 | 0
  PsyDO - Hypomania, mild | 1 | 0
  PsyDO - Hypomania, moderate | 0 | 0
  PsyDO - Hypomania, severe | 0 | 0
  PsyDO - Intentional self-injury, mild | 1 | 0
  PsyDO - Intentional self-injury, moderate | 0 | 0
  PsyDO - Intentional self-injury, severe | 0 | 0
  PsyDO - Libido decreased, mild | 1 | 0
  PsyDO - Libido decreased, moderate | 0 | 0
  PsyDO - Libido decreased, severe | 0 | 0
  PsyDO - Nightmare, mild | 0 | 0
  PsyDO - Nightmare, moderate | 0 | 1
  PsyDO - Nightmare, severe | 0 | 0
  General Disorders (GD) - Any Event, mild | 10 | 16
  GD - Any Event, moderate | 5 | 5
  GD - Any Event, severe | 0 | 0
  GD - Drug Withdrawal Syndrome, mild | 2 | 6
  GD - Drug Withdrawal Syndrome, moderate | 2 | 3
  GD - Drug Withdrawal Syndrome, severe | 0 | 0
  GD - Thirst, mild | 4 | 9
  GD - Thirst, moderate | 0 | 0
  GD - Thirst, severe | 0 | 0
  GD - Malaise, mild | 1 | 1
  GD - Malaise, moderate | 2 | 0
  GD - Malaise, severe | 0 | 0
  GD - Feeling abnormal, mild | 0 | 1
  GD - Feeling abnormal, moderate | 0 | 1
  GD - Feeling abnormal, severe | 0 | 0
  GD - Irritability, mild | 0 | 0
  GD - Irritability, moderate | 1 | 1
  GD - Irritability, severe | 0 | 0
  GD - Chills, mild | 1 | 0
  GD - Chills, moderate | 0 | 0
  GD - Chills, severe | 0 | 0
  GD - Edema, mild | 1 | 0
  GD - Edema, moderate | 0 | 0
  GD - Edema, severe | 0 | 0
  GD - Edema peripheral, mild | 1 | 0
  GD - Edema peripheral, moderate | 0 | 0
  GD - Edema peripheral, severe | 0 | 0
  GD - Pain, mild | 1 | 0
  GD - Pain, moderate | 0 | 0
  GD - Pain, severe | 0 | 0
  Skin & tissue disorders (SDO) - Any Event, mild | 6 | 8
  SDO - Any Event, moderate | 1 | 6
  SDO - Any Event, severe | 0 | 1
  SDO - Urticaria, mild | 0 | 1
  SDO - Urticaria, moderate | 0 | 4
  SDO - Urticaria, severe | 0 | 0
  SDO - Rash, mild | 1 | 2
  SDO - Rash, moderate | 0 | 1
  SDO - Rash, severe | 0 | 0
  SDO - Eczema, mild | 1 | 1
  SDO - Eczema, moderate | 0 | 0
  SDO - Eczema, severe | 0 | 0
  SDO - Hyperhidrosis, mild | 2 | 0
  SDO - Hyperhidrosis, moderate | 0 | 0
  SDO - Hyperhidrosis, severe | 0 | 0
  SDO - Hypoesthesia facial, mild | 0 | 2
  SDO - Hypoesthesia facial, moderate | 0 | 0
  SDO - Hypoesthesia facial, severe | 0 | 0
  SDO - Pruritus generalised, mild | 0 | 1
  SDO - Pruritus generalised, moderate | 0 | 1
  SDO - Pruritus generalised, severe | 0 | 0
  SDO - Alopecia, mild | 0 | 0
  SDO - Alopecia, moderate | 0 | 1
  SDO - Alopecia, severe | 0 | 0
  SDO - Alopecia areata, mild | 0 | 1
  SDO - Alopecia areata, moderate | 0 | 0
  SDO - Alopecia areata, severe | 0 | 0
  SDO - Dermatitis Contact, mild | 0 | 0
  SDO - Dermatitis Contact, moderate | 1 | 0
  SDO - Dermatitis Contact, severe | 0 | 0
  SDO - Erythema, mild | 1 | 0
  SDO - Erythema, moderate | 0 | 0
  SDO - Erythema, severe | 0 | 0
  SDO - Hemorrhage subcutaneous, mild | 0 | 0
  SDO - Hemorrhage subcutaneous, moderate | 0 | 0
  SDO - Hemorrhage subcutaneous, severe | 0 | 1
  SDO - Hyperkeratosis, mild | 0 | 1
  SDO - Hyperkeratosis, moderate | 0 | 0
  SDO - Hyperkeratosis, severe | 0 | 0
  SDO - Pigmentation disorder, mild | 1 | 0
  SDO - Pigmentation disorder, moderate | 0 | 0
  SDO - Pigmentation disorder, severe | 0 | 0
  SDO - Sweat Gland Disorder, mild | 0 | 1
  SDO - Sweat Gland Disorder, moderate | 0 | 0
  SDO - Sweat Gland Disorder, severe | 0 | 0
  Investigations (INV) - Any Event, mild | 5 | 10
  INV - Any Event, moderate | 1 | 2
  INV - Any Event, severe | 0 | 0
  INV - Alanine Aminotransferase increased, mild | 3 | 4
  INV - Alanine Aminotransferase increased, moderate | 0 | 0
  INV - Alanine Aminotransferase increased, severe | 0 | 0
  INV - Weight decreased, mild | 0 | 3
  INV - Weight decreased, moderate | 0 | 0
  INV - Weight decreased, severe | 0 | 0
  INV - Aspartate Aminotransferase increased, mild | 0 | 2
  INV-Aspartate Aminotransferase increased, moderate | 0 | 0
  INV - Aspartate Aminotransferase increased, severe | 0 | 0
  INV - Blood Bilirubin increased, mild | 1 | 1
  INV - Blood Bilirubin increased, moderate | 0 | 0
  INV - Blood Bilirubin increased, severe | 0 | 0
  INV - Glucose urine present, mild | 0 | 1
  INV - Glucose urine present, moderate | 0 | 1
  INV - Glucose urine present, severe | 0 | 0
  INV - Protein urine present, mild | 0 | 2
  INV - Protein urine present, moderate | 0 | 0
  INV - Protein urine present, severe | 0 | 0
  INV - White Blood Cell Count decreased, mild | 0 | 1
  INV - White Blood Cell Count decreased, moderate | 0 | 1
  INV - White Blood Cell Count decreased, severe | 0 | 0
  INV - Blood pressure decreased, mild | 0 | 0
  INV - Blood pressure decreased, moderate | 1 | 0
  INV - Blood pressure decreased, severe | 0 | 0
  INV - Electrocardiogram T wave inversion, mild | 1 | 0
  INV - Electrocardiogram T wave inversion, moderate | 0 | 0
  INV - Electrocardiogram T wave inversion, severe | 0 | 0
  INV - Hematocrit decreased, mild | 0 | 1
  INV - Hematocrit decreased, moderate | 0 | 0
  INV - Hematocrit decreased, severe | 0 | 0
  INV - Hemoglobin decreased, mild | 0 | 1
  INV - Hemoglobin decreased, moderate | 0 | 0
  INV - Hemoglobin decreased, severe | 0 | 0
  INV - Red Blood Cell Count decreased, mild | 0 | 1
  INV - Red Blood Cell Count decreased, moderate | 0 | 0
  INV - Red Blood Cell Count decreased, severe | 0 | 0
  Musculoskeletal Disorders (MD) - Any Event, mild | 9 | 6
  MD - Any Event, moderate | 0 | 2
  MD - Any Event, severe | 0 | 0
  MD - Back Pain, mild | 1 | 1
  MD - Back Pain, moderate | 0 | 2
  MD - Back Pain, severe | 0 | 0
  MD - Musculoskeletal stiffness, mild | 3 | 1
  MD - Musculoskeletal stiffness, moderate | 0 | 0
  MD - Musculoskeletal stiffness, severe | 0 | 0
  MD - Myalgia, mild | 2 | 1
  MD - Myalgia, moderate | 0 | 0
  MD - Myalgia, severe | 0 | 0
  MD - Neck Pain, mild | 0 | 2
  MD - Neck Pain, moderate | 0 | 0
  MD - Neck Pain, severe | 0 | 0
  MD - Pain in extremity, mild | 2 | 0
  MD - Pain in extremity, moderate | 0 | 0
  MD - Pain in extremity, severe | 0 | 0
  MD - Arthralgia, mild | 0 | 1
  MD - Arthralgia, moderate | 0 | 0
  MD - Arthralgia, severe | 0 | 0
  MD - Fasciitis, mild | 1 | 0
  MD - Fasciitis, moderate | 0 | 0
  MD - Fasciitis, severe | 0 | 0
  Respiratory Disorders (RTM) - Any Event, mild | 4 | 6
  RTM -Any Event, moderate | 0 | 3
  RTM -Any Event, severe | 0 | 0
  RTM - Upper respiratory Tract inflammation, mild | 3 | 3
  RTM-Upp. respiratory Tract inflammation, moderate | 0 | 1
  RTM-Upp. respiratory Tract inflammation, severe | 0 | 0
  RTM - Asthma, mild | 0 | 2
  RTM - Asthma, moderate | 0 | 1
  RTM - Asthma, severe | 0 | 0
  RTM - Cough, mild | 0 | 1
  RTM - Cough, moderate | 0 | 1
  RTM - Cough, severe | 0 | 0
  RTM - Pharyngolaryngeal Pain, mild | 1 | 0
  RTM - Pharyngolaryngeal Pain, moderate | 0 | 0
  RTM - Pharyngolaryngeal Pain, severe | 0 | 0
  Injury and complications (IPPC) - Any Event, mild | 2 | 2
  IPPC - Any Event, moderate | 1 | 3
  IPPC - Any Event, severe | 0 | 0
  IPPC - Contusion, mild | 0 | 2
  IPPC - Contusion, moderate | 0 | 0
  IPPC - Contusion, severe | 0 | 0
  IPPC - Intentional Overdose, mild | 1 | 0
  IPPC - Intentional Overdose, moderate | 0 | 1
  IPPC - Intentional Overdose, severe | 0 | 0
  IPPC - Head Injury, mild | 0 | 0
  IPPC - Head Injury, moderate | 0 | 1
  IPPC - Head Injury, severe | 0 | 0
  IPPC - Joint sprain, mild | 0 | 1
  IPPC - Joint sprain, moderate | 0 | 0
  IPPC - Joint sprain, severe | 0 | 0
  IPPC - Rib fracture, mild | 0 | 0
  IPPC - Rib fracture, moderate | 1 | 0
  IPPC - Rib fracture, severe | 0 | 0
  IPPC - Thermal Burn, mild | 0 | 0
  IPPC - Thermal Burn, moderate | 0 | 1
  IPPC - Thermal Burn, severe | 0 | 0
  IPPC - Wound, mild | 1 | 0
  IPPC - Wound, moderate | 0 | 0
  IPPC - Wound, severe | 0 | 0
  Ear Disorders (ED) - Any Event, mild | 3 | 2
  ED - Any Event, moderate | 0 | 0
  ED - Any Event, severe | 0 | 0
  ED - Tinnitus, mild | 2 | 2
  ED - Tinnitus, moderate | 0 | 0
  ED - Tinnitus, severe | 0 | 0
  ED - Ear Discomfort, mild | 1 | 0
  ED - Ear Discomfort, moderate | 0 | 0
  ED - Ear Discomfort, severe | 0 | 0
  Eye Disorders (EyeDO) - Any Event, mild | 0 | 1
  EyeDO - Any Event, moderate | 0 | 3
  EyeDO - Any Event, severe | 0 | 0
  EyeDO - Chalazion, mild | 0 | 0
  EyeDO - Chalazion, moderate | 0 | 2
  EyeDO - Chalazion, severe | 0 | 0
  EyeDO - Abnormal sensations in eye, mild | 0 | 0
  EyeDO - Abnormal sensations in eye, moderate | 0 | 1
  EyeDO - Abnormal sensations in eye, severe | 0 | 0
  EyeDO - Conjunctival haemorrhage, mild | 0 | 1
  EyeDO - Conjunctival haemorrhage, moderate | 0 | 0
  EyeDO - Conjunctival haemorrhage, severe | 0 | 0
  Metabolism Disorders (MetDO) - Any Event, mild | 2 | 1
  MetDO - Any Event, moderate | 1 | 0
  MetDO - Any Event, severe | 0 | 0
  MetDO - Anorexia, mild | 0 | 1
  MetDO - Anorexia, moderate | 1 | 0
  MetDO - Anorexia, severe | 0 | 0
  MetDO - Dehydration, mild | 2 | 0
  MetDO - Dehydration, moderate | 0 | 0
  MetDO - Dehydration, severe | 0 | 0
  MetDO - Hyperlipidemia, mild | 1 | 0
  MetDO - Hyperlipidemia, moderate | 0 | 0
  MetDO - Hyperlipidemia, severe | 0 | 0
  MetDO - Hypovitaminosis, mild | 1 | 0
  MetDO - Hypovitaminosis, moderate | 0 | 0
  MetDO - Hypovitaminosis, severe | 0 | 0
  Vascular Disorders (VD) - Any Event, mild | 2 | 2
  VD - Any Event, moderate | 0 | 0
  VD - Any Event, severe | 0 | 0
  VD - Hot Flush, mild | 1 | 2
  VD - Hot Flush, moderate | 0 | 0
  VD - Hot Flush, severe | 0 | 0
  VD - Hypertension, mild | 1 | 0
  VD - Hypertension, moderate | 0 | 0
  VD - Hypertension, severe | 0 | 0
  Blood & Lymph Disorders (BLD) - Any Event, mild | 0 | 2
  BLD - Any Event, moderate | 0 | 1
  BLD - Any Event, severe | 0 | 0
  BLD - Anemia, mild | 0 | 1
  BLD - Anemia, moderate | 0 | 1
  BLD - Anemia, severe | 0 | 0
  BLD - Lymphadenopathy, mild | 0 | 1
  BLD - Lymphadenopathy, moderate | 0 | 0
  BLD - Lymphadenopathy, severe | 0 | 0
  Hepatobiliary disorders (HD) - Any Event, mild | 1 | 1
  HD - Any Event, moderate | 0 | 1
  HD - Any Event, severe | 0 | 0
  HD - Hepatic Function abnormal, mild | 1 | 1
  HD - Hepatic Function abnormal, moderate | 0 | 1
  HD - Hepatic Function abnormal, severe | 0 | 0
  Reproductive Disorders (RBD) - Any Event, mild | 0 | 1
  RBD - Any Event, moderate | 0 | 1
  RBD - Any Event, severe | 0 | 1
  RBD - Galactorrhea, mild | 0 | 0
  RBD - Galactorrhea, moderate | 0 | 1
  RBD - Galactorrhea, severe | 0 | 0
  RBD - Menometrorrhagia, mild | 0 | 1
  RBD - Menometrorrhagia, moderate | 0 | 0
  RBD - Menometrorrhagia, severe | 0 | 0
  RBD - Premenstrual Syndrome, mild | 0 | 0
  RBD - Premenstrual Syndrome, moderate | 0 | 0
  RBD - Premenstrual Syndrome, severe | 0 | 1
  Cardiac Disorders (CD) - Any Event, mild | 1 | 1
  CD - Any Event, moderate | 0 | 0
  CD - Any Event, severe | 0 | 0
  CD - Palpitations, mild | 1 | 1
  CD - Palpitations, moderate | 0 | 0
  CD - Palpitations, severe | 0 | 0
  Renal & Urinary Disorders (RUD) - Any Event, mild | 0 | 2
  RUD - Any Event, moderate | 0 | 0
  RUD - Any Event, severe | 0 | 0
  RUD - Dysuria, mild | 0 | 1
  RUD - Dysuria, moderate | 0 | 0
  RUD - Dysuria, severe | 0 | 0
  RUD - Pollakiuria, mild | 0 | 1
  RUD - Pollakiuria, moderate | 0 | 0
  RUD - Pollakiuria, severe | 0 | 0
  Endocrine Disorders (ENDO) - Any Event, mild | 0 | 1
  ENDO - Any Event, moderate | 0 | 0
  ENDO - Any Event, severe | 0 | 0
  ENDO - Hyperprolactinaemia, mild | 0 | 1
  ENDO - Hyperprolactinaemia, moderate | 0 | 0
  ENDO - Hyperprolactinaemia, severe | 0 | 0

ADVERSE EVENTS:
Arm/Group | Placebo | Bupropion SR
Serious Adverse Events (participants affected / at risk) | 0 | 5
Other Adverse Events (participants affected / at risk) | 124/159 | 125/166
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Placebo | Bupropion SR
Depressed level of Consciousness (Nervous system disorders) | 0/159 | 2/166
Convulsion (Nervous system disorders) | 0/159 | 1/166
Bipolar Disorder (Psychiatric disorders) | 0/159 | 1/166
Mania (Psychiatric disorders) | 0/159 | 1/166
Asthma (Respiratory, thoracic and mediastinal disorders) | 0/159 | 1/166
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=159) | Bupropion SR (N=166)
Nasopharyngitis (Infections and infestations) | 31 | 28
Nausea (Gastrointestinal disorders) | 21 | 26
Depression (Psychiatric disorders) | 20 | 14
Dizziness (Nervous system disorders) | 16 | 16
Somnolence (Psychiatric disorders) | 10 | 8
Headache (Nervous system disorders) | 9 | 15
Diarrhea (Gastrointestinal disorders) | 9 | 7
Vomiting (Gastrointestinal disorders) | 8 | 7
Drug Withdrawal syndrome (General disorders) | 4 | 9
Thirst (General disorders) | 4 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the Publication of results from all centers of a multi-center trial but requests that reports based on Single-site data not precede the primary publication of the entire clinical trial.